CLINICAL TRIAL: NCT07008261
Title: Prospective Evaluation of Robot-assisted Cystectomies With Regard to Blood Loss, Pain and Transfusion Requirements.
Brief Title: Robot-assisted Cystectomies With Regard to Blood Loss, Pain and Transfusions.
Status: Recruiting | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Armin N. Flinspach, senior physician, Goethe University
Other Study IDs: PBM in robot cystectomies
Record Dates: First submitted 2025-05-27; First posted 2025-06-06 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-06

CONDITIONS: Transfusions; Cystectomy; Blood Loss Requiring Transfusion; Anaemia; Anaemia Postoperative; Pain, Postoperative
MeSH Terms: conditions — Anemia; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robot assistet: Robot assistet laparoscopic cystectomy
- Conventional: Conventional laparotomy for cystektomie

SUMMARY:
What influence does robot-assisted surgical treatment in the sense of a radical cystectomy and possibly bladder reconstruction have on blood loss, pain and transfusion requirements? We intend to conduct a corresponding prospective observational study at a tertiary centre.

ELIGIBILITY:
Inclusion Criteria:

* planned radical cystectomy

Exclusion Criteria:

* ASA classification V
* Previously known coagulation disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a mostly oncological indication for radical cystectomy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
perioperative blood loss | 6 hours
  perioperative blood loss

SECONDARY OUTCOMES:
Preoperative iron deficiency | up to 4 weeks prior surgery
  Preoperative messured iron deficiency
RBC transfusion | perioperative up to hospital discharge or death (up to 4 weeks)
  Number of RBC transfusions

CONTACTS AND LOCATIONS:
Locations (1):
- Uniklinikum, Frankfurt am Main, Germany